CLINICAL TRIAL: NCT03760822
Title: Second-Line Chemotherapy With Ramucirumab +/- Paclitaxel in Elderly Advanced Gastric or Gastroesophageal Junction Cancer Patients
Acronym: SOCRATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 55 - SOCRATE
Record Dates: First submitted 2018-07-17; First posted 2018-11-30 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Stomach Cancer; Stomach Neoplasm; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: ramucirumab; elderly patient; second line therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramucirumab (Experimental): IV ramucirumab at 8 mg/kg on D1 and D15
  Interventions: Drug: Ramucirumab
- Ramucirumab + Paclitaxel (Active Comparator): IV ramucirumab at 8 mg/kg on D1 and D15 IV paclitaxel at 80 mg/m² on D1, D8 and D15
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — IV ramucirumab at 8 mg/kg on D1 and D15
  Other Names: Cyramza
Drug: Paclitaxel — IV paclitaxel at 80 mg/m² on D1, D8 and D15
  Other Names: Abraxane
  Arms: Ramucirumab + Paclitaxel

SUMMARY:
The primary objective is to evaluate six months survival rate and quality of life at 4 months of ramucirumab alone or in combination with paclitaxel in patients aged 70 years or more who have stomach or GEJ adenocarcinoma and whose first line of fluoropyrimidine- and platinumcontaining treatment has failed.

The co-primary endpoints are the following:

* Six months survival rate
* Quality of life at 4 months as assessed by the following three target dimensions of the EORTC QLQ-ELD14 questionnaire: mobility, illness burden and worries about the future

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable, locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma, whatever HER2 status
* Aged ≥ 70 years
* WHO < 2
* Estimated life expectancy > 3 months
* Measurable or non-measurable disease according to RECIST 1.1 criteria
* Documented progression during first-line fluoropyrimidine- and platinum- or irinotecan containing chemotherapy (with or without anthracycline), or during the 4 months following the last cycle of such chemotherapy administered for metastatic or locally advanced disease, or during the 6 months following the last dose of adjuvant therapy containing fluoropyrimidine and platinium (treatment by immunotherapy is allowed)
* Adequate hepatic, renal and hematologic function:

  * ANC ≥ 1 500 / mm3, platelets ≥ 100 000 / mm3, hemoglobin ≥ 9 g/dL
  * Blood creatinine ≤ 1.5 x ULN and creatinine clearance (MDRD formula) ≥ 40 mL/min
  * Total bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 3 x ULN (≤ 5 x ULN if hepatic metastasis)
  * INR ≤ 1.5 or INR ≤ 3 for patients taking AVK and PTT ≤ 5 seconds above the ULN
  * Dipstick proteinuria ≤ 1+ or 24 hour proteinuria < 1 g in total
* EORTC QLQ-C30 + QLQ-ELD14, completed and faxed to the Randomization, Management and Analysis Center of the FFCD
* IADL geriatric questionnaire, completed and faxed to Randomization Management and Analysis Center of FFCD
* Signed informed consent

Exclusion Criteria:

* Known cerebral metastasis
* Prior treatment by taxanes
* Prior treatment with an antiangiogenic
* Neuropathy of grade ≥ 2 (NCI-CTCAE 4.0)
* Unresolved partial or total bowel obstruction, inflammatory bowel disease (such as Crohn's disease or ulcerative colitis) or extensive gastrointestinal (GI) resection combined with chronic diarrhea
* GI perforation and/or fistulae in the 6 months preceding randomization.
* GI bleeding within the last 3 months of grade ≥ 3 (NCI-CTCAE 4.0)
* Chronic use of antiplatelet drugs (including aspirin, but a daily intake of ≤ 325 mg/day is accepted), non-steroidal anti-inflammatory drugs (ibuprofen, naproxen), dipyridamole, clopidogrel or similar agents
* Any arterial thromboembolic event (such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack) in the 6 months preceding randomization
* A life-threatening episode of pulmonary embolism in the 6 months preceding randomization
* Deep-vein thrombosis, pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant" during the 3 months prior to first dose of protocol therapy
* Uncompensated congestive heart failure or uncontrolled arrhythmia
* Uncontrolled hypertension (≥ 140/90 mm Hg for > 4 weeks) despite properly observed antihypertensive therapy
* Cirrhosis at a level of Chilg-Pugh B or C; or cirrhosis (any degree) with a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Serious or unhealed wound, peptic ulcer or fracture within 28 days of randomization
* Radiotherapy or major surgery within 28 days of prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior the first dose of protocol therapy
* Known allergy to paclitaxel or ramucirumab
* Another concomitant cancer or a history of cancer in the last 5 years, except cervical carcinoma in situ, cutaneous basal-cell or squamous-cell carcinoma, or any other carcinoma in situ deemed to be successfully treated
* Lack of effective contraception in patients (man and/or women) of childbearing age, and/or their
* Persons deprived of liberty or under supervision
* Impossibility of undergoing medical monitoring during the trial for geographic, social or psychological reasons

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient survival rate at 6 months | at 6 months
  Rate of patients alive
Quality of life at 4 months as assessed by the following dimension of the EORTC QLQ-ELD14 questionnaire: mobility | at 4 months
  Derived from items 31,33 and 34of the ELD14 questionnaire. The score is from 0 to 100. The endpoint is defined as the difference of at least 10 points (clinical significance) between baseline score and 4-months score.
Quality of life at 4 months as assessed by the following dimension of the EORTC QLQ-ELD14 questionnaire: worries about the future | at 4 months
  Derived from items 31,33 and 34of the ELD14 questionnaire. The score is from 0 to 100. The endpoint is defined as the difference of at least 10 points (clinical significance) between baseline score and 4-months score.
Quality of life at 4 months as assessed by the following dimension of the EORTC QLQ-ELD14 questionnaire: illness burden | at 4 months
  Derived from items 43 and 44of the ELD14 questionnaire. The score is from 0 to 100. The endpoint is defined as the difference of at least 10 points (clinical significance) between baseline score and 4-months score

SECONDARY OUTCOMES:
Overall survival | 6 months
  Defined as time to death (whatever cause is) or for patients alive time to last news.
Time to treatment failure | 6 months
  Time between randomization and disease progression, treatment interruption or death
Progression-free survival | 6 months
  Progression-free survival (clinical and/or radiological) determined by the investigator based on RECIST V1.1

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Lièvre, Pr, Principal Investigator — CHU de Pontchaillou - Rennes
Locations (38):
- France (38):
  - CH -, Abbeville
  - CH - Albi, Albi
  - PRIVEE - L'Europe, Amiens
  - CAC - ICO Site Paul Papin, Angers
  - Privee - Hopital Prive, Antony
  - Ch - Victor Dupouy, Argenteuil
  - Ch - Metz Thionville Mercy, Ars-Laquenexy
  - Ch - Ght Unyon Auxerre, Auxerre
  - Privee - Institut Du Cancer Avignon Provence, Avignon
  - Ch - Cote Basque, Bayonne
  - Ch - Beauvais Ch, Beauvais
  - Chu - Jean Minjoz, Besançon
  - Privee - Tivoli, Bordeaux
  - PRIVEE - Polyclinique Saint Privat, Boujan-sur-Libron
  - Ch - Duchenne, Boulogne-sur-Mer
  - Ch - Pierre Oudot, Bourgoin
  - Privee - Pasteur Lanroze, Brest
  - Cac - François Baclesse, Caen
  - Chu - Côte de Nacre, Caen
  - Ch - Jean Rougier, Cahors
  - Privee - Infirmerie Protestante, Caluire-et-Cuire
  - CH -, Carcassonne
  - Ch - Castres Mazamet Chi, Castres
  - Prive - Médipole de Savoie, Challes-les-Eaux
  - Prive - Sainte Marie, Chalon-sur-Saône
  - CH -, Cholet
  - Ch - Hopitaux Civils de Colmar, Colmar
  - Hopitaux civils de Colmar, Colmar
  - Chu - Louis Mourier, Colombes
  - Prive - Saint Côme, Compiègne
  - Prive - Cédres, Cornebarrieu
  - Chu - Henri Mondor, Créteil
  - Prive - Centre Leonard de Vinci, Dechy
  - Cac - Gf Leclerc, Dijon
  - Chu - Francois Mitterrand, Dijon
  - CH -, Dunkirk
  - CHI - Elbeuf Louviers Val de Reuil, Elbeuf
  - Clinique privée - CENTRE CARIO, Plérin

IPD SHARING:
Plan to Share IPD: Undecided